



## **CONSENT FORM**

Study title: Objective response detection to natural speech stimuli for optimisation of hearing aid fitting evaluation

Researcher name: Dr Frederique J Vanheusden, Dr Katie Ireland, Constantina Georga

ERGO number: 30123

Please initial the box(es) if you agree with the statement(s):

| I have read and understood the information sheet (Version 1.0, 15/08/2017) and have had the opportunity to ask questions about the study. |
|---|
| I understand my participation is voluntary and I may withdraw (at any time) for any reason without my rights being affected. |
| I agree that my anonymised data will be made available at the secured data repository of the University of Southampton for inclusion in future research studies and could be distributed to third parties in accordance to the University's legal standards. I am aware that I can ask to have my data withdrawn from the repository at any time during or after the study |
| Research can sometimes find out important information about my hearing function. I give permission for the research team to give advice about possible issues with my hearing and which steps I could take to avoid further hearing dysfunction. |
| I agree to take part in this research project and agree for my data to be used for the purpose of this study. |
| Name of participant (print name) |
| Signature of participant |
| Date |
| Name of researcher (print name) |
| Signature of researcher |
| Date |